CLINICAL TRIAL: NCT02211144
Title: Safety and Pharmacokinetics of BIRB 796 BS Tablets Administered Twice Daily Orally (Total Daily Dose 90, 120, 150 or 180 mg) to Healthy Human Subjects for 14 Days. A Placebo-controlled, Dose Escalation Study Double Blinded at Each Dose Level
Brief Title: Safety and Pharmacokinetics of BIRB 796 BS Tablets Administered Twice Daily Orally to Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1175.21
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BIRB 796 BS (Experimental): in escalating doses
  Interventions: Drug: BIBR 796 BS; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBR 796 BS
  Arms: BIRB 796 BS
Drug: Placebo

SUMMARY:
Study to assess the safety and pharmacokinetics of BIRB 796 BS tablets administered as multiple daily doses at various dose levels

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Female subjects who were not lactating and not of child bearing potential as defined by surgically sterile or post menopausal (no periods for at least 12 months and elevated follicle stimulating hormone (FSH) with low estradiol while on no estrogen supplementation). Females were to use barrier contraception (e.g. condoms) prior to administration of study medication, during the study and at least one month after release from the study. Women must have had negative blood pregnancy tests
* Age ≥ 18 and ≤ 60 years
* Body mass index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
* Able to communicate well with the investigator and to comply with study requirements
* Laboratory values within a clinically defined reference range

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate, and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* History of vasculitis (past history of fever, malaise, myalgias, rash, etc.)
* Intake of drugs with a long half-life (> 24 hours) (< 1 month prior to administration or during the trial)
* Use of any drugs, which might influence the results of the trial, (< 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (< 1 months prior to administration (at least 10 times the relevant elimination half-life) or during the trial)
* Having had prescription medication 2 weeks prior to study drug administration or over the counter medication 1 week prior to study drug administration (at least 10 times the relevant elimination half-life)
* Smoker
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Use of methylxanthine-containing drinks or foods (coffee, tea, cola, energy drinks, chocolate, etc.), grapefruit or grapefruit juice, alcohol, green tea, or tobacco < 5 days prior to administration of study drug
* Blood donation or loss > 400 mL (< 1 month prior to administration or during the trial)
* Excessive physical activities (< 5 days prior to administration or during the trial)
* Following specific laboratory findings: white blood cell count, C-reactive protein, gamma-glutamyl-transferase, aspartate transaminase, alanine transaminase, or glutamate dehydrogenase above the normal range; any erythrocytes or > 15 mg/dl protein on urine dipstick if not menstruating
* Any EKG value outside of the reference range of clinical relevance including, but not limited to QTcB > 480 ms or QRS interval > 110 ms
* History of any familial bleeding disorder
* Inability to comply with dietary regimen of study centre
* Inability to comply with investigator's instructions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2002-03; Primary Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant changes in vital signs (pulse rate, systolic and diastolic blood pressure) | up to day 21
Number of patients with clinically relevant changes in laboratory parameters | up to day 21
Number of patients with clinical relevant findings in electrocardiogram (ECG) | up to day 21
Number of patients with adverse events | up to 35 days
Clinical assessment of tolerability on a 4-point scale | day 21

SECONDARY OUTCOMES:
Maximum observed plasma concentration during steady state dosing interval (Cmax,ss) | up to day 16
area under the plasma concentration versus time curve at different time points (AUC) | up to day 16
Time to the maximum plasma concentration at steady state (tmax,ss) | up to day 16
Elimination half-life (t1/2) | up to day 16
Terminal elimination rate constant (λz) | up to day 16
Average steady state plasma concentration (Css) | up to day 16
Mean residence time (MRT) | up to day 16
Total apparent oral clearance of drug from plasma after oral administration (CL/F ) | up to day 16
Apparent volume of distribution based on terminal elimination phase, divided by F (bioavailability factor) (Vz/F) | up to day 16
Morning trough plasma concentration prior day 14 | on day 2, 3, 5, 7, 9, 13 and 14